CLINICAL TRIAL: NCT00643552
Title: Muscle Strength, Physical Work Capacity and Functional Performance in Individuals With Down Syndrome
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Lori Ploutz-Snyder, Syracuse University
Other Study IDs: 4973
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Down Syndrome
Keywords: Muscle Strength
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will evaluate muscle strength and its relationship to everyday function in individuals with Down Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Down Syndrome
* Mild or moderate mental retardation
* Able to tolerate exercise testing

Exclusion Criteria:

* Uncontrolled cardiovascular disease
* orthopedic limitations to exercise

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)